CLINICAL TRIAL: NCT05692037
Title: Yttrium-90 Carbon Microspheres in Patients With Unresectable Colorectal Liver Metastases: A Multicentre, Prospective, Open-label, Single-arm Trial
Brief Title: Yttrium-90 Carbon Microspheres in Patients With Unresectable Colorectal Liver Metastases
Acronym: NRT-uCRLM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Dean, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANCE2303-NRT6003
Record Dates: First submitted 2022-12-25; First posted 2023-01-20 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Unresectable Colorectal Liver Metastases
MeSH Terms: interventions — Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yttrium-90 carbon microspheres (Experimental): Single dose of yttrium-90 carbon microspheres injection. Patients will be assessed by SPECT-CT imaging within 24 hours for yttrium-90 distribution in the chest and upper abdomen, including extrahepatic shunts, intrahepatic distribution, and target lesion distribution as expected.Ten Patients will be tested for the radioactivity of yttrium-90 in blood, urine, and feces (if available).
  Interventions: Combination Product: Selective internal radiation therapy (SIRT) with yttrium-90 carbon microspheres

INTERVENTIONS:
Combination Product: Selective internal radiation therapy (SIRT) with yttrium-90 carbon microspheres — Yttrium-90 carbon microspheres SIRT

SUMMARY:
To evaluate the efficacy and safety of yttrium-90 carbon microspheres in patients with unresectable colorectal liver metastases

DETAILED DESCRIPTION:
The efficacy and safety of yttrium-90 carbon microspheres in patients with unresectable colorectal liver metastases remain unknown. This multicentre, prospective, open-label, single-arm trial is designed to evaluate the safety and efficacy of yttrium-90 carbon microspheres in patients with unresectable colorectal liver metastases. The primary endpoints are the progression-free survival rates of liver target lesions. While the secondary endpoints include the safety, tumor control, and the distribution characteristics of yttrium-90 carbon microspheres.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group performance status ≤ 1;
2. Expected survival time ≥ 3 months;
3. Confirmed liver metastasis of colorectal cancer;
4. Complete resection and no local recurrence of the primary colorectal cancer;
5. Intolerance, failure to the previous anti-tumor treatments or, or recurrence liver metastasis after surgical resection;
6. Without extrahepatic metastases, inoperable or refuse surgical resection;
7. At least one well defined tumor (RECIST 1.1);
8. Tumor burden ≤ 50% of the total liver volume;
9. Child-Pugh score ≤ 7;
10. Adequate organ function: ① Blood routine [no blood transfusion or colony-stimulating factor (G-CSF) treatment within 14 days]: absolute neutrophil count ≥ 1.5 × 109/L; platelet ≥ 75 × 109/L; hemoglobin ≥ 90 g/L; ② Liver function: total bilirubin ≤ 2 times upper limit of normal (ULN); alanine transaminase and aspartate aminotransferase ≤ 5. 0 ULN; alkaline phosphatase ≤ 2.5 ULN; Albumin > 30 g/L; ③ Renal function: Cr ≤ 1.5 ULN; creatinine clearance ≥ 50 mL/min (calculated according to Cockcroft-Gault formula); ④ Coagulation function: international normalized ratio, prothrombin time and activated partial thromboplastin time were less than 1.5 ULN; ⑤ Cardiovascular function: left ventricular ejection fraction ≥ 50%;
11. According to CTCAE 5.0 standard, all adverse events of previous systematic anti-cancer treatment have recovered to baseline or ≤ 1 grade, [except for the following: neuropathy induced by previous anti-cancer treatment is stable (≤ 2 grade) and hair loss];
12. Women and men of childbearing age must agree to take strict and effective contraceptive measures during the study period and within 6 m after the end of the trial. Men are forbidden to donate sperm. The pregnancy test results of female patients of childbearing age during the screening period and within 24 hours before administration must be negative.

Exclusion Criteria:

1. With previous history of hepatic encephalopathy;
2. Severe pulmonary insufficiency (forced expiratory volume at one second / forced vital capacity < 50% or forced expiratory volume at one second /predicting value < 50% or maximum volume per minute < 50 L/min);Obvious chronic obstructive pulmonary disease or interstitial pneumonia;
3. Percentage of hepatopulmonary shunt > 10%, or the single lung radiation absorbed dose > 30 Gy;
4. With hepatic artery malformation and unable to intubate hepatic artery;
5. Tumor thrombus in main portal vein;
6. Have received radiotherapy or transcatheter arterial chemoembolization (patients who have received transcatheter arterial non-iodized oil chemoembolization are judged by researchers);
7. The last anti-tumor treatment (surgery, chemotherapy, immunotherapy, targeted therapy) was less than 4 weeks before the drug administration;
8. Clinical manifestations of portal hypertension, moderate-severe or refractory ascites, or decompensated liver cirrhosis;
9. Major surgery or severe trauma within 28 days before yttrium-90 administration;
10. Participated in other trial within 1 month before yttrium-90 administration;
11. Pregnant and lactating women;
12. Serious infections in active stage or need systematic treatment;
13. With positive results of HIV antibody test;
14. The researchers judge that there is unresolved toxicity from previous treatment and will continue to exist, which may endanger the safety of patients;
15. The researcher judged clinical or laboratory examination abnormality or other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Rate of Liver Target Lesions | 3 months after yttrium-90 injection
  Survival probability of patients without imaging progression of liver target lesions

SECONDARY OUTCOMES:
Adverse events | Up to 24 months
  Rate of adverse events
Yttrium-90 distribution | Within 24 hours
  Assessed by SPECT-CT imaging in the chest and upper abdomen, including extrahepatic shunts, intrahepatic distribution, and target lesion distribution as expected.Ten Patients will be tested for the radioactivity of yttrium-90 in blood, urine, and feces (if available)
Objective response rate (ORR) | Up to 24 months
  Evaluated by the investigator and independent image review committee respectively (CTCAE 1.1)
Duration of response (DOR) | Up to 24 months
  Time without imaging progression, evaluated by the investigator and independent image review committee respectively (CTCAE 1.1)
Hepatic progression-free survival (hPFS) | Up to 24 months
  Time without imaging progression of liver target lesions, evaluated by the investigator and independent image review committee respectively (CTCAE 1.1)
Time to progression (TTP) | Up to 24 months
  Time with tumor progression, evaluated by the investigator and independent image review committee respectively (CTCAE 1.1)
Progression-free survival (PFS) | Up to 24 months
  Evaluated by the investigator and independent image review committee respectively (CTCAE 1.1)
Overall survival (OS) | Up to 24 months
  Survival time
Disease control rate (DCR) | Up to 24 months
  Probability of tumor control

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No